CLINICAL TRIAL: NCT00250068
Title: Phase II Study of Aerosolized Liposomal 9-Nitro-20 (S)- Camptothecin (L9NC)
Brief Title: Study of Aerosolized Liposomal 9-Nitro-20 (S)- Camptothecin (L9NC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Claire F Verschraegen, MD; Principal Investigator, University of New Mexico
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1402C
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2008-10

CONDITIONS: Lung Diseases; Cancer
Keywords: Phase II; Aerosol Delivery; NSCLC; 9-Nitrocamptothecin
MeSH Terms: conditions — Lung Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Liposomal 9-Nitrocamptothecin — Dose: 0.4 mg/ml of 9-NC in aerosol reservoir for 60 minutes (= daily dose of 0.52 mg/m2/day) per day X5 every week, X8 weeks, then observe for 2 weeks. One course = 10 weeks

SUMMARY:
To determine the overall response rate to liposomal 9-Nitro-20 (S)-Camptothecin (L9NC) administered by aerosolization in patients with non-small-cell lung cancer (any stage.

To determine toxicity profile of L9NC administered by aerosolization for 5 consecutive days per week X 8 weeks, every 10 weeks.

To perform a pharmacology study of L9NC in the plasma, and the lungs after aerosolization. A specific protocol will be written for this part.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized Phase II trial of DLPC-9NC administered by aerosol 5 consecutive days per week for 8 weeks every 10 weeks.

Dose: 0.4 mg/ml of 9-NC in aerosol reservoir for 60 minutes (= daily dose of 0.52 mg/m2/day) per day X5 every week, X8 weeks, then observe for 2 weeks. One course = 10 weeks.

Patients that have a resectable lung cancer will only receive one course of treatment and will be operated on about two weeks after completing the 8-week course.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years of age or older, with resectable lung cancer (any stage) or stage 3b, 4, or recurrent, nonresectable, non-small-cell lung carcinoma, who have failed standard chemotherapy or radiotherapy for their disease or who refuse standard therapy are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of >1,500 or cells/mm3 and platelet count >100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.
* Patients must not have a known symptomatic respiratory disease other than cancer, and must have a pulmonary function test equal to >50% FEV1, >50% FEV1/FVC, >50% TLC, and >50% DLCO of predicted values.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Any criteria that is borderline and may lead to ineligibility will be reviewed by the PI, who may override the eligibility criteria, after receiving sponsor agreement, if entry into the study is deemed to potentially benefit the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine the overall response rate to liposomal 9-Nitro-20 (S)-Camptothecin (L9NC) administered by aerosolization in patients with non-small-cell lung cancer (any stage). | disease progression or unacceptable toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Claire F Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States